CLINICAL TRIAL: NCT02083601
Title: Caring for Caregivers: Supporting Caregivers of Youth With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erin Hayes Kelly, PhD (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor-Investigator, Erin Hayes Kelly, PhD, Principal Investigator, Shriners Hospitals for Children
Organization: Shriners Hospitals for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 288993
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Spinal Cord Injuries
Keywords: Caregivers; Spinal Cord Injuries; Psychology, Educational; Counseling; Outcome Assessment (Health Care)
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychological Support (Experimental): The intervention group will participate in the 2-day, in-person Parent Forum and receive monthly phone calls from a mental health professional for 12 months.
  Interventions: Behavioral: Parent Forum; Behavioral: Psychological support
- No Psychological Support (Other): This comparison group will attend the 2-day, in-person Parent Forum but will not receive long-term psychological support.
  Interventions: Behavioral: Parent Forum

INTERVENTIONS:
Behavioral: Parent Forum — In-person psychoeducational workshop that provides education (including problem-solving training) and psychological/peer support for caregivers of youth with SCI.
Behavioral: Psychological support — Outreach from a mental health professional in the form of monthly phone calls for 12 months.
  Arms: Psychological Support

SUMMARY:
The current study will implement and evaluate a multi-component, psychoeducational intervention for caregivers of children with spinal cord injury (SCI) ages 7-12. Two hypotheses will be tested. First, caregivers who participate in the intervention group will demonstrate better outcomes than caregivers in the control group. Second, children with SCI whose caregivers participate in the intervention group will demonstrate better outcomes than children with SCI whose caregivers participate in the control group.

DETAILED DESCRIPTION:
The primary objective of this study is to implement and evaluate an intervention for caregivers of children with spinal cord injury (SCI) ages 7-12. A further objective of this pilot study is to identify which outcomes are being affected by the intervention. Past research has highlighted psychoeducational intervention (i.e., interventions including both educational/skills-building components and psychological support) as most effective in terms of impacting caregiver functioning. The current study will recruit 44 caregivers and their children with SCI. All caregivers will participate in a 2-day Parent Forum, an in-person educational session. Caregivers will then be randomly assigned to receive monthly phone calls from a mental health professional ("intervention group") or no additional targeted support ("control group"). We expect that caregivers who participate in the intervention group and their children will demonstrate better outcomes than caregivers in the control group and their children.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregivers of youth with SCI ages 7-12 years.
* Youth sustained their SCI at least one year ago.
* Both the caregiver and child are able to speak English.
* Both the caregiver and child are able and willing to sign informed consent/assent and Health Insurance Portability and Accountability Act (HIPAA) compliant research authorization.

Exclusion Criteria:

* Caregiver or child has significant cognitive limitations and/or psychiatric comorbidities. These conditions will be identified by a clinical psychologist or physician.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Longitudinal changes in Social Problem Solving Inventory-Revised (SPSI-R) over time | Baseline, Immediately after Parent Forum, 6 months, 12 months, 18 months
  This short-form will be completed by parents to assess their social problem solving skills. There are four subscales: positive and negative problem orientation, rational problem solving, impulsivity/carelessness style, and avoidance style.
Longitudinal changes in Satisfaction with Life Scale (SWLS) over time | Baseline, 6 months, 12 months, 18 months
  This self-report measure will be used to assess subjective life satisfaction or QOL among caregivers.
Longitudinal changes in Hospital Anxiety and Depression Scale (HADS) over time | Baseline, 6 months, 12 months, 18 months
  This self-report measure will be used to assess depression, anxiety, and emotional distress.
Longitudinal changes in Social support/Social integration questions over time | Baseline, 6 months, 12 months, 18 months
  Consistent with past research, caregivers will be asked about their satisfaction with social support, and the number of relatives, friends, neighbors, and others that they see or hear from at least once each month, feel close to, or feel they can call on for help with things like chores or transportation.
Longitudinal changes in Caregiver Burden Interview over time | Baseline, 6 months, 12 months, 18 months
  A modified version of the brief 12- item version of the Caregiver Burden Interview will be administered to caregivers. Originally developed for caregivers of cognitively impaired older adults, this survey will be adapted for parents of children with SCI.
Longitudinal changes in Medical Outcomes Study Short Form Health Survey (SF-36) over time | Baseline, 6 months, 12 months, 18 months
  This self-report measure will be used to assess caregivers' health perceptions and general well-being. The SF-36 including the following scales: physical functioning, physical role functioning, pain, general health, energy/fatigue, social functioning, and emotional role functioning and mental health.
Longitudinal changes in Revised Scale for Caregiving Self-Efficacy over time | Baseline, Immediately after Parent Forum, 6 months, 12 months, 18 months
  A modified version of this self-report scale will be used to assess the belief that the caregiver has about his or her ability to successfully carry out certain kinds of behaviors. This measure includes 15 items within 3 subscales: self-efficacy for obtaining respite, responding to disruptive patient behaviors, and controlling upsetting thoughts about caregiving. Originally created for caregivers of cognitively impaired older adults, this survey will also be adapted for parents of children with SCI.
Longitudinal changes in Physical Health Form over time | Baseline, 6 months, 12 months, 18 months
  This survey was developed by the current research team and will be completed by the caregiver about their child's bowel and bladder incontinence and the presence of pressure ulcers.
Longitudinal changes in Pediatric Quality of Life Inventory (PedsQL) over time | Baseline, 6 months, 12 months, 18 months
  Caregivers will complete the proxy-report versions of the general core scales to assess four areas of their child's health-related QOL: physical, emotional, social, and school functioning. Children will complete the self-report general core scales to assess four areas of their health-related QOL: physical, emotional, social, and school functioning.
Evaluation tool to assess intervention satisfaction over time | Immediately after Parent Forum, 6 months, 12 months, 18 months
  Caregivers will be asked about their satisfaction with the intervention components (including resulting peer relationships), including the Parent Forum (for all caregivers) and outreach from the mental health professional (for caregivers in the intervention group only).
Longitudinal changes in Faces Pain Scale/Visual Analog Scale over time | Baseline, 6 months, 12 months, 18 months
  These 10-point pain scales will be used to assess pain intensity in youth ages 7-8 and 9-12, respectively. These children will be asked about pain intensity at the time of survey completion (acute pain).
Longitudinal changes in Children's Depression Inventory: Second Edition-Short Form (CDI-2-SF) over time | Baseline, 6 months, 12 months, 18 months
  The short form of this self-report measure yields an overall depression score and will be administered to children ages 7-12.
Longitudinal changes in Revised Children's Manifest Anxiety Scale: Second Edition-Short Form (RCMAS-2-SF) over time | Baseline, 6 months, 12 months, 18 months
  The short form of this self-report measure is designed to assess the level and nature of anxiety with subscales assessing physiological anxiety, worry, social anxiety, defensiveness, and inconsistent responding. The RCMAS-2-SF will be administered to children ages 7-12.

CONTACTS AND LOCATIONS:
Overall Officials: Erin H Kelly, PhD, Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Chicago, Illinois, United States